CLINICAL TRIAL: NCT07001241
Title: Effects of a Telehealth Exercise Program for Rural Cancer Survivors With Cancer-related Fatigue Including Integrated Longitudinal Assessments of Objective Physical Function and Fatty Acid Oxidation
Brief Title: Telehealth Exercise Program Evaluating Fatigue and Physical Function in Rural Cancer Survivors
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 24-1398.cc; R01CA292482 (NIH)
Record Dates: First submitted 2025-05-23; First posted 2025-06-03 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Cancer-related Fatigue; Breast Cancer; Prostate Cancer
Keywords: Prostate Cancer; Exercise; Telehealth; Breast Cancer; Metabolism; Physical function
MeSH Terms: conditions — Breast Neoplasms; Prostatic Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Participants are randomized to an intervention group or wait-list control group. Participants in both groups complete all study assessments (primary outcomes). Following all study assessments with no intervention, participants in the wait-list control group will receive the full exercise program.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Telehealth Exercise Program (Experimental): The BfitBwell-TP (Telehealth Program) intervention is designed specifically for rural cancer survivors with cancer-related fatigue (CRF). It is personalized to each participant, addresses known barriers to exercise participation in rural survivors, and incorporates the experience and infrastructure of the established clinical BfitBwell Cancer Exercise Program. BfitBwell-TP is delivered completely via existing and accessible telehealth technologies including: videoconference sessions with a cancer exercise specialist, exercise programming and text communication using a personal training smartphone/internet application, and emailed surveys. CRF is assessed throughout the program with additional telehealth sessions initiated if it does not improve as predicted based on a reference chart developed with BfitBwell data.
  Interventions: Behavioral: Telehealth Exercise Program
- Waitlist Control Group (No Intervention): This group will be instructed to not change their current physical activity and exercise routines while completing all study assessments (including brief assessments every two weeks). After completing a final assessment following the 12-week wait period, they will receive the full exercise intervention (see Experimental Arm for description).

INTERVENTIONS:
Behavioral: Telehealth Exercise Program — BfitBwell-TP is a 12-week telehealth exercise intervention. Exercise prescriptions are created, personalized, and delivered by Cancer Exercise Specialists. Exercise content is delivered using a combination of videoconference sessions and a commercial personal training application (accessible via smartphone or internet browser). Patient-reported symptoms (specifically cancer-related fatigue) are assessed every two weeks via emailed surveys. Survey scores are compared to a reference chart of predicted improvements during the program, developed from an established clinical exercise oncology program. Additional videoconference sessions are initiated for participants demonstrating lower than expected symptom improvement, with the goal of adapting the current exercise prescription to improve symptom response.
  Other Names: BfitBwell Telehealth Program (BfitBwell-TP)
  Arms: Telehealth Exercise Program

SUMMARY:
This study investigates the efficacy of a telehealth exercise program designed specifically for rural cancer survivors with cancer-related fatigue (CRF). Small dried blood samples and measures of physical function will be collected throughout the program. The main questions it aims to answer are:

* Does the exercise program improve CRF in rural cancer survivors?
* How do CRF, metabolism, and physical function change during the exercise program? Researchers will compare the program to a wait-list control group. This group will complete all study measures without without changing current physical activity before receiving the full exercise program.

Participants will:

* Complete a virtual physical assessment before and after the program.
* Complete brief virtual assessments and collect dried blood samples (at home and mailed in) every two weeks during the program.
* Receive a personalized exercise program including virtual sessions and remote exercise programming with a cancer exercise specialist (after a 12-week wait period in the wait-list control group).
* Optional: Willing participants will visit a study site for a laboratory-based exercise assessment before and after the program.

DETAILED DESCRIPTION:
This study investigates the efficacy of a telehealth exercise program designed specifically for rural cancer survivors with cancer-related fatigue (CRF). The 12-week program is designed to be delivered completely via remote methods including: telehealth exercise sessions with cancer exercise specialists, additional exercise programming delivered through a personal training smartphone/internet application, and regular symptom monitoring via emailed surveys. Symptoms (CRF) are plotted against a reference chart of anticipated changes during the program, with additional telehealth sessions initiated if symptoms do not improve as predicted. Program efficacy is investigated using a randomized controlled trial with a wait-list control group (N=134, Aim 1). The control group will receive the exercise program following a 12-week wait period.

Possible mechanisms of action are assessed throughout the program (every two weeks) using accessible methods (Aim 2). Fatty acid oxidation is measured via dried blood spots collected remoted and mailed to the primary study site. Physical function is measured via brief telehealth assessments.

Changes in molecular responses to acute exercise and changes in body composition will be explored in a controlled laboratory assessment in participants able and willing to travel to participating sites (N=40, Aim 3). Small blood samples are collected before and after a standardized treadmill exercise session. Body composition is measured non-invasively in a small chamber using air displacement. This laboratory assessment occurs before and after the program (or wait period).

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 and < 90 years of age. 2. Diagnosis of breast or prostate cancer. 3. Cancer treatment criteria: 3a. Completion of treatment with curative intent > 3 months prior to and < 5 years from study initiation.

3b. Treatment must include hormonal, radiation, chemotherapy, and/or immunotherapy. Those who have received only surgery are not eligible.

3c. Individuals diagnosed with breast cancer currently receiving maintenance hormonal therapy, with no planned treatment changes in the next six months, are eligible.

4. Home zip code meeting Health Resources & Services Administration (HRSA) definition of rural (data.hrsa.gov/tools/rural-health).

5. Presence of at least moderate fatigue (>3/10 per National Comprehensive Cancer Network guidelines).

6. Access to high-speed home internet. 7. Possession of smartphone or laptop with front-facing camera. 8. Capable and willing to give informed consent. 9. Willing to participate in a 12-week telehealth exercise intervention or 12-week waiting period prior to intervention with brief remote physical assessments and dried blood spot collection every 2 weeks.

10. Able and willing to provide contact information for a local support individual to assist with any possible adverse events.

11. Able and willing to provide contact information for a local primary care provider to address medical issues potentially arising during study activities.

12. Able to provide signed physician clearance for exercise if indicated by the Physical Activity Readiness Questionnaire (PAR-Q+) or National Comprehensive Cancer Network exercise safety screening questions.

Exclusion Criteria:

1. Eastern Cooperative Oncology Group (ECOG) Performance Status Grade ≥ 2.
2. Current or planned cancer-related treatments (except maintenance hormonal therapies) in the next six months.

2a. For individuals with a prostate cancer diagnosis, those currently receiving androgen deprivation therapy (ADT), or those who have previously received ≥ 12 months of ADT, are not eligible.

3. Plans to relocate to a non-rural location in the next six months. 4. Presence of a disease or condition that affects the ability of an individual to safely participate in an exercise intervention (e.g. recent cardiac event or chronic obstructive pulmonary disease).

4a. These conditions are identified in the PAR-Q+. 5. Presence or history of metabolic disease (e.g. diabetes or uncontrolled hyper- or hypothyroidism).

5a. Participants with pre-diabetes, metabolic syndrome, or diabetes managed with metformin only will be eligible, with this variable tracked for later analysis.

6. Current participation in another exercise oncology program.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2025-10-08 (Actual); Primary Completion 2028-08 (Estimated); Study Completion 2030-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline in FACIT-Fatigue (cancer-related fatigue) score at Week 12 | Baseline, Week 12
  The Functional Assessment of Chronic Illness Therapy - Fatigue scale (FACIT-Fatigue) is a common standardized measure of cancer-related fatigue. It contains 13 items with total score ranging from 0 to 52, with higher scores indicating less fatigue.

SECONDARY OUTCOMES:
Change from Baseline in FACIT-Fatigue (cancer-related fatigue) score at Week 24 | Baseline, Week 24
  The Functional Assessment of Chronic Illness Therapy - Fatigue scale (FACIT-Fatigue) is a common standardized measure of cancer-related fatigue. It contains 13 items with total score ranging from 0 to 52, with higher scores indicating less fatigue.
Change from Baseline in FACT-G (quality of life) score at Week 12 | Baseline, Week 12
  The Functional Assessment of Cancer Treatment - General scale (FACTG-G) is a common standardized measure of quality of life in cancer survivors. It contains 27 items with total score ranging from 0 to 108, with higher scores indicating better quality of life.
Pattern of change in FACIT-Fatigue (cancer-related fatigue) score during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  The Functional Assessment of Chronic Illness Therapy - Fatigue scale (FACIT-Fatigue) is a common standardized measure of cancer-related fatigue. It contains 13 items with total score ranging from 0 to 52, with higher scores indicating less fatigue.
  Scores will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.
Change from Baseline in FACT-G (quality of life) score at Week 24 | Baseline, Week 24
  The Functional Assessment of Cancer Treatment - General scale (FACTG-G) is a common standardized measure of quality of life in cancer survivors. It contains 27 items with total score ranging from 0 to 108, with higher scores indicating better quality of life.
Change from Baseline in HADS (anxiety and depression) scores at Week 12 | Baseline, Week 12
  The Hospital Anxiety and Depression Scale (HADS) is a common standardized measure of anxiety and depression in clinical populations. It contains 14 items yielding Anxiety and Depression scores. Scores range from 0 to 21, with higher scores indicating more anxiety or depressive symptoms.
Change from Baseline in HADS (anxiety and depression) scores at Week 24 | Baseline, Week 24
  The Hospital Anxiety and Depression Scale (HADS) is a common standardized measure of anxiety and depression in clinical populations. It contains 14 items yielding Anxiety and Depression scores. Scores range from 0 to 21, with higher scores indicating more anxiety or depressive symptoms.
Change from Baseline in EORTC QLQ-FA12 (cancer-related fatigue) scores at Week 12 | Baseline, Week 12
  The European Organisation for Research and Treatment of Cancer Group Quality of Life Questionnaire Fatigue 12 (EORTC QLQ-FA12) is a recently developed measure of cancer-related fatigue with multiple subscales (physical fatigue, emotional fatigue, and cognitive fatigue). It contains 12 items, with scores ranging from 0 to 100, and higher scores indicating higher fatigue symptoms.
Change from Baseline in EORTC QLQ-FA12 (cancer-related fatigue) scores at Week 24 | Baseline, Week 24
  The European Organisation for Research and Treatment of Cancer Group Quality of Life Questionnaire Fatigue 12 (EORTC QLQ-FA12) is a recently developed measure of cancer-related fatigue with multiple subscales (physical fatigue, emotional fatigue, and cognitive fatigue). It contains 12 items, with scores ranging from 0 to 100, and higher scores indicating higher fatigue symptoms.
Change from Baseline in 2MST (physical function) at Week 12 | Baseline, Week 12
  The Two-Minute Step Test (2MST) is a submaximal test of aerobic capacity. Participants step in place for two minutes, raining each knee to a pre-specified height. Final measure is number of steps performed, with more steps indicating higher aerobic capacity.
Change from Baseline in CS (physical function) at Week 12 | Baseline, Week 12
  The Chair Stand Test (CS) is an assessment of lower extremity function and muscular strength. Participants move from a seated position to standing and back as many times as possible in 30 s. Final measure is number of completed stands, with more stands indicating higher muscular strength and function.
Change from Baseline in GS (physical function) at Week 12 | Baseline, Week 12
  Gait Speed (GS) is a common clinical measure of physical function. Participants are timed while walking at a 'usual' pace for 4 m. Final measure is m/s, with faster speeds indicating higher function.
Change from Baseline in TUG (physical function) at Week 12 | Baseline, Week 12
  The Timed Up and Go test (TUG) is a common clinical measure of physical function. Participants are timed while standing from a chair, walking 3 m, turning around, and returning to sit in the chair. Final measure is time to perform, with lower times indicating higher function.
Change from Baseline in SLB (physical function) at Week 12 | Baseline, Week 12
  Single Leg Balance (SLB) is a common clinical measure of balance and physical function. Participants are timed while standing on one leg with no external support (for up to 30 s). Final measure is time able to balance, with higher times indicating higher function.
Change from Baseline in daily physical activity (PA) at Week 12 | Baseline, Week 12
  Daily physical activity will be assessed for a 7-day period and calculated as average steps/day. This will be collected with a study provided commercial activity tracker.
Change from Baseline in average sleep time at Week 12 | Baseline, Week 12
  Sleep time, assessed as time in bed at night, will be assessed over a 7-day period and averaged. This will be measured with a study provided commercial fitness tracker.
Change from Baseline in fatty acid oxidation at Week 12 | Baseline, Week 12
  Fatty acid oxidation will be calculated as the ratio of medium- to long-chain acylcarnitines in metabolomic and lipidomic data acquired from high-throughput liquid chromatography-mass spectrometry. Samples are collected remotely as dried blood spots and mailed to the primary study site.
Change from Baseline in dynamic exercise metabolic profiles at Week 12 | Baseline, Week 12
  This measure is optional and performed at a participating study site. Small blood samples are collected before, after, and 30 min after a standard 36 min moderate intensity treadmill walking session. Dynamic metabolic profiles will be investigated by comparing analyses from the different timepoints (e.g. before-to-after exercise, recovery from after-to-30 minutes after exercise, etc.), using metabolomic and lipidomic data acquired from the collected samples via high-throughput liquid chromatography-mass spectrometry.
Change from Baseline in body composition at Week 12 | Baseline, Week 12
  This measure is optional, performed during assessments at a participating study site. Body composition is measured while participants sit in a small, closed chamber for approximately two minutes, via air displacement plethysmography. The measure is presented as percent fat mass and percent lean mass.
Pattern of change in FACT-G (quality of life) score during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  The Functional Assessment of Cancer Treatment - General scale (FACTG-G) is a common standardized measure of quality of life in cancer survivors. It contains 27 items with total score ranging from 0 to 108, with higher scores indicating better quality of life.
  Scores will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.
Pattern of change in HADS (anxiety and depression) scores during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  The Hospital Anxiety and Depression Scale (HADS) is a common standardized measure of anxiety and depression in clinical populations. It contains 14 items yielding Anxiety and Depression scores. Scores range from 0 to 21, with higher scores indicating more anxiety or depressive symptoms.
  Scores will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.
Pattern of change in EORTC QLQ-FA12 (cancer-related fatigue) scores during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  The European Organisation for Research and Treatment of Cancer Group Quality of Life Questionnaire Fatigue 12 (EORTC QLQ-FA12) is a recently developed measure of cancer-related fatigue with multiple subscales (physical fatigue, emotional fatigue, and cognitive fatigue). It contains 12 items, with scores ranging from 0 to 100, and higher scores indicating higher fatigue symptoms.
  Scores will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.
Pattern of change in 2MST (physical function) during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  The Two-Minute Step Test (2MST) is a submaximal test of aerobic capacity. Participants step in place for two minutes, raining each knee to a pre-specified height. Final measure is number of steps performed, with more steps indicating higher aerobic capacity.
  Measure will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.
Pattern of change in CS (physical function) during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  The Chair Stand Test (CS) is an assessment of lower extremity function and muscular strength. Participants move from a seated position to standing and back as many times as possible in 30 s. Final measure is number of completed stands, with more stands indicating higher muscular strength and function.
  Measure will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.
Pattern of change in GS (physical function) during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  Gait Speed (GS) is a common clinical measure of physical function. Participants are timed while walking at a 'usual' pace for 4 m. Final measure is m/s, with faster speeds indicating higher function.
  Measure will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.
Pattern of change in TUG (physical function) during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  The Timed Up and Go test (TUG) is a common clinical measure of physical function. Participants are timed while standing from a chair, walking 3 m, turning around, and returning to sit in the chair. Final measure is time to perform, with lower times indicating higher function.
  Measure will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.
Pattern of change in SLB (physical function) during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  Single Leg Balance (SLB) is a common clinical measure of balance and physical function. Participants are timed while standing on one leg with no external support (for up to 30 s). Final measure is time able to balance, with higher times indicating higher function.
  Measure will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.
Pattern of change in fatty acid oxidation during exercise intervention or wait period | Baseline, Week 2, Week 4, Week 6, Week 8, Week 10, Week 12
  Fatty acid oxidation will be calculated as the ratio of medium- to long-chain acylcarnitines in metabolomic and lipidomic data acquired from high-throughput liquid chromatography-mass spectrometry. Samples are collected remotely as dried blood spots and mailed to the primary study site.
  Measure will be collected every two weeks during the intervention (or wait period) and change patterns established as the changes between adjacent timepoints.

CONTACTS AND LOCATIONS:
Overall Officials: Ryan J Marker, PhD, DPT, Principal Investigator — University of Colorado, Denver
Locations (2):
- United States (2):
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - University of Montana, Missoula, Montana

IPD SHARING:
Plan to Share IPD: Yes
De-identified research outcomes data and protocols will be made upon request, at the study PI's discretion.
Supporting Information: Study Protocol, ICF, Analytic Code
Time Frame: Following publication of major investigation findings (approximately 2030) through required data storage (approximately 2037).
Access Criteria: De-identified research data will be made available, upon request, following the publication of major investigation findings. Data will be stored on University of Colorado servers, and user registration will be required to access the data, in accordance with NIH Data Sharing Policy Guidelines. An agreement to the following conditions will be required: 1) data may only be used for research purposes, 2) no attempt will be made to identify research participants, 3) data will be destroyed following analysis completion, and 4) data will not be distributed to third parties. Access to data will be identified in all publications to maintain wide availability to the research community in accordance with University policies and the NIH Principles and Guidelines document.